CLINICAL TRIAL: NCT01922414
Title: Laser Versus Ultrasonic Lithotripsy in Percutaneous Nephrolithotomy for Staghorn Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Assistant Professor of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Staghorn Laser; Staghorn Laser vs US (Other: Urology and Nephrology Center)
Record Dates: First submitted 2013-08-01; First posted 2013-08-14 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Stones
Keywords: Staghorn stones; Percutaneous nephrolithotomy; Laser; Randomized trial; Lithotripsy
MeSH Terms: conditions — Kidney Calculi | interventions — Lasers; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser (Active Comparator): Patients will undergo Laser lithotripsy
  Interventions: Device: Laser
- Ultrasonic (Active Comparator): Patients will undergo ultrasonic lithotripsy
  Interventions: Device: Ultrasonic

INTERVENTIONS:
Device: Laser — Patients will undergo laser lithotripsy durin PNL
  Arms: Laser
Device: Ultrasonic — Patients will undergo ultrasonic lithotripsy during PNL
  Arms: Ultrasonic

SUMMARY:
This study will be conducted to compare the results of Laser and ultrasonic lithotripsy in disintegration of staghorn stones during percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
Patients with complete staghorn stones who are eligible to percutaneous nephrolithotomy (PNL) will be randomized between two groups.

Group 1: will undergo Laser lithotripsy during PNL Group 2: will undergo ultrasonic lithotripsy during PNL

ELIGIBILITY:
Inclusion Criteria:

1. Complete staghorn stones (filling the renal pelvis and branching to 3 major calyces
2. Age: 18-70 years

Exclusion Criteria:

1. Congenital renal anomalies such as horse shoe kidney.
2. Contraindications to PNL such as bleeding tendency and uncontrolled hypertension.
3. Associated pathological features requiring open intervention such as UPJO
4. Partial staghorn stones (filling the renal pelvis and branching to 2 major calyces)
5. Giant staghorn stone (very large staghorn stone that branch and re-branch in hugely dilated calyceal system)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Stone Free rate | Patients will be followed for 3 months after the procedure
  Assessment of stone free rate after 3 months from treatment using NCCT

SECONDARY OUTCOMES:
Assessment of the safety of each technique | From the start of the operation till 3 months after discharge from the hospital
  Measurement of complication rates, classifications of the severity of complications
Operative time | An expected average of 3 hours
  Measurement of the time from start of ureteral catheter fixation till the fixation of the nephrostomy tube
Hospital stay | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R. EL-Nahas, MD, Principal Investigator — faculty of medicine
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakhlia, Egypt

REFERENCES:
- [Background] Preminger GM, Assimos DG, Lingeman JE, Nakada SY, Pearle MS, Wolf JS Jr; AUA Nephrolithiasis Guideline Panel). Chapter 1: AUA guideline on management of staghorn calculi: diagnosis and treatment recommendations. J Urol. 2005 Jun;173(6):1991-2000. doi: 10.1097/01.ju.0000161171.67806.2a. No abstract available. PMID 15879803
- [Background] Bagley DH. Expanding role of ureteroscopy and laser lithotripsy for treatment of proximal ureteral and intrarenal calculi. Curr Opin Urol. 2002 Jul;12(4):277-80. doi: 10.1097/00042307-200207000-00003. PMID 12072646
- [Background] Jou YC, Shen JH, Cheng MC, Lin CT, Chen PC. Percutaneous nephrolithotomy with holmium: Yttrium-aluminum-garnet laser and fiber guider--report of 349 cases. Urology. 2005 Mar;65(3):454-8. doi: 10.1016/j.urology.2004.09.069. PMID 15780354
- [Background] Gu Z, Qi J, Shen H, Liu J, Chen J. Percutaneous nephroscopic with holmium laser and ultrasound lithotripsy for complicated renal calculi. Lasers Med Sci. 2010 Jul;25(4):577-80. doi: 10.1007/s10103-010-0769-x. Epub 2010 Mar 16. PMID 20232221
- [Background] Mandal S, Goel A, Goyal NK. Re: Staghorn morphometry: a new tool for clinical classification and prediction model for percutaneous nephrolithotomy monotherapy. (From: Mishra S, Sabnis RB, Desai M. J Endourol 2012;26:6-14). J Endourol. 2012 Aug;26(8):1099. doi: 10.1089/end.2012.0088. Epub 2012 Apr 17. No abstract available. PMID 22509933
- [Background] Qi S, Li L, Liu R, Qiao B, Zhang Z, Xu Y. Impact of stone branch number on outcomes of percutaneous nephrolithotomy for treatment of staghorn calculi. J Endourol. 2014 Feb;28(2):152-7. doi: 10.1089/end.2013.0333. Epub 2013 Nov 20. PMID 24083829
- [Background] el-Nahas AR, Eraky I, Shokeir AA, Shoma AM, el-Assmy AM, el-Tabey NA, Soliman S, Elshal AM, el-Kappany HA, el-Kenawy MR. Factors affecting stone-free rate and complications of percutaneous nephrolithotomy for treatment of staghorn stone. Urology. 2012 Jun;79(6):1236-41. doi: 10.1016/j.urology.2012.01.026. Epub 2012 Apr 1. PMID 22465085
- [Background] Desai M, De Lisa A, Turna B, Rioja J, Walfridsson H, D'Addessi A, Wong C, Rosette On Behalf Of The Croes Pcnl Study Group J. The clinical research office of the endourological society percutaneous nephrolithotomy global study: staghorn versus nonstaghorn stones. J Endourol. 2011 Aug;25(8):1263-8. doi: 10.1089/end.2011.0055. Epub 2011 Jul 20. PMID 21774666
- [Result] Jou YC, Shen CH, Cheng MC, Lin CT, Chen PC. High-power holmium:yttrium-aluminum-garnet laser for percutaneous treatment of large renal stones. Urology. 2007 Jan;69(1):22-5; discussion 25-6. doi: 10.1016/j.urology.2006.08.1114. PMID 17270603
- [Result] Sun Y, Gao X, Zhou T, Chen S, Wang L, Xu C, Hou J. 70 W holmium: yttrium-aluminum-garnet laser in percutaneous nephrolithotomy for staghorn calculi. J Endourol. 2009 Oct;23(10):1687-91. doi: 10.1089/end.2009.1536. PMID 19732015
- [Result] Malik HA, Tipu SA, Mohayuddin N, Sultan G, Hussain M, Hashmi A, Naqvi SA, Rizvi SA. Comparison of holmium: Yag laser and pneumatic lithoclast in percutaneous nephrolithotomy. J Pak Med Assoc. 2007 Aug;57(8):385-7. PMID 17902519
- [Result] El-Nahas AR, Eraky I, Shokeir AA, Shoma AM, El-Assmy AM, El-Tabey NA, El-Kappany HA, El-Kenawy MR. Long-term results of percutaneous nephrolithotomy for treatment of staghorn stones. BJU Int. 2011 Sep;108(5):750-4. doi: 10.1111/j.1464-410X.2010.09942.x. Epub 2010 Dec 16. PMID 21166763